CLINICAL TRIAL: NCT00931333
Title: Non Comparative, Monocentric, Prospective, Phase II, Study of Calcium Phosphate Cement MCPC Efficacy and Safety for Bone Filling in Vertebral Site
Brief Title: Efficacy and Safety Study of Non-percutaneous Vertebroplasty With Macroporous Calcium Phosphate Cement (MCPC)
Acronym: VERTEBRO-MCPC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2009/03
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Vertebra Trauma
Keywords: Vertebroplasty; spine; vertebra height; adverse events; calcium phosphate bone cement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: non percutaneous vertebroplasty

INTERVENTIONS:
Procedure: non percutaneous vertebroplasty — The patient will undergo general anaesthetic. With a low invasive approach, 4 screws will be placed in pedicles of vertebra under and above the fractured vertebra. The reduction of the fracture will be realised by a smooth movement, and screws positions will be verified by a radio control, with a guided navigation system. The stems will be placed and locked. After the screw positioning, the fractured vertebra pedicles will be reached by a low invasive approach, using a 6 mm trocar, to raise, if necessary, the vertebral plate. Then the cement will be injected in the vertebral body, under radio control. When the maximal volume (6 to 8 ml) is reached, or if an extra vertebral leak is detected, the cement injection is stopped. Then the incision is closed. The next day, the patient will be placed in a corset for a 2 months period.

SUMMARY:
The macroporous calcium phosphate cement, MCPC, which composition is close to bone, is malleable and biocompatible, and has intrinsic radio opacity and good ability to undergo mechanical constraints. After the filling of the bone cavity, the cement hardens. Interestingly, this calcium phosphate cement has no exothermic hardening (on the contrary, the ordinary cements used nowadays cause necrotic lesions in tissues around during this phase) and favours vascularisation, cellular colonisation and bone healing. Thanks to its resorbability, the MCPC cement is replaced little by little by a physiologic bone. This last property is very important for young people needing a vertebroplasty after a traumatism.

Thus, it will be tested in a low-invasive surgery, a non-percutaneous vertebroplasty, consisting in filling with the MCPC the body of the broken vertebra, after its stabilization thanks to 4 interpedicular screws. This protocol will be proposed to patients 1 to 3 weeks after the trauma having caused the fracture.

The follow up will last 12 months with 5 visits (2 days, and 3, 4, 6 and 12 months after vertebroplasty), 2 CT scanners before inclusion and at 12 months, 2 EOS (ultra low dose imager replacing classical radiography) at 5 and 12 months, questionnaires (visual analogic scale for pain, and quality of life with OSWESTRY and SF36 scales) before inclusion and at 2 days, and 3, 4, 6 and 12 months, and biological exams (CRP/VS, for inflammation) at each visit except 2 days after surgery. An osteodensitometry will be performed at 3 months.

DETAILED DESCRIPTION:
The macroporous calcium phosphate cement, MCPC, which composition is closer to bone than acrylic cement, is malleable and biocompatible, and has intrinsic radio opacity and good biomechanical properties (12 +/- 3 Mpa in 24 hours). After the filling of the bone cavity, the cement hardens in situ thanks to hydrolysis and apatite precipitation. Interestingly, this calcium phosphate cement has no exothermic hardening (on the contrary, the PMMA causes necrotic lesions in tissues around during this phase). During the dissolution, a macroporosity takes form between biphasic calcium phosphate granules. That permits vascularisation, cellular colonisation and bone healing. Thanks to its resorbability, the MCPC cement is replaced by a physiologic tissue. This last property is very important for young people needing a vertebroplasty after a traumatism.

The issue is to validate this biomaterial with appropriate mechanical, biocompatibility properties and intrinsic radio opacity, and that can favour bone regeneration, with a lower frequency of leak and risk enhancement of other vertebra fracture. The MCPC will thus be tested on few patients to assess its efficacy and security for bone filling in vertebra site.

Thus, it will be used in a low-invasive surgery, a non-percutaneous vertebroplasty, consisting in filling with the MCPC the body of the broken vertebra, after its stabilization thanks to 4 interpedicular screws. This protocol will be proposed to 21 patients 1 to 3 weeks after the trauma having caused the fracture. The follow up will last 12 months with 5 visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years old, BMI < 30
* Stable and important fracture of the vertebral body between T9 and L5
* Diagnostic maximum 3 weeks after the trauma causing the fracture
* Type A1 to A3 (MAGERL scale) assessed by CT scan
* Lumbar local traumatic angle > 10°, and thoracic > 15°
* Given informed consent
* Patient with French health system

Exclusion Criteria:

* For women: no efficient contraception (intra uterine device, or contraceptive pill)
* Pregnant or feeding women
* Fractures due to metastasis or multiple myeloma
* Symptomatic compression of the spinal cord
* Multi site vertebroplasty
* Scoliosis with a Cobb angle > 20°
* Surgery zone local infection
* All surgical contraindications
* Immune system abnormalities, immune deficiency or suppression, HIV or BHV or CHV (positive serology)
* Severe hyperparathyroidism: calcium > 2,45 mmol/l and [PTH] ≥ 50pg / ml
* Uncontrolled diabetes (untreated or non stabilized by treatment)
* Long corticoid treatment (more than 6 months and stopped since less than 3 months)
* Chemotherapy
* All contra indication to MCPC: osteomyelitis, bone degenerative disease or necrosis of surgery site.
* Known allergy to indigotine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The efficiency of non-percutaneous vertebroplasty using MCPC, in 18 to 65 years old patients, after a huge trauma, will be evaluated based on evaluation of the vertebra height by measuring local traumatic angle. | At the 4th month after the surgical procedure

SECONDARY OUTCOMES:
The proportion of Severe Adverse Events frequency (cement leak, new fractures, late huge loss of vertebra height) and inflammatory response | before inclusion and at 3 months, 4 months, 5 months, 12 months
Pain intensity: difference between before inclusion and during follow up. Evaluation with Visual Analogic Scale. | before inclusion and at 2 days, and 3, 4, 6 and 12 months
Quality of life: difference between before inclusion and during follow up. Evaluation with OSWESTRY and SF 36 scales. | before inclusion and at 2 days, and 3, 4, 6 and 12 months.
The evolution of bone formation and MCPC resorption: quantification of bone reconstruction. | CT scan at 6 and 12 months after surgery, and with osteodensitometry at 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles LE HUEC, Professor, Principal Investigator — University Hospital Bordeaux, France; Antoine BENARD, MD, Study Chair — University Hospital Bordeaux, France
Locations (1):
- Service d'orthopédie-traumatolologie (C), Hôpital Pellegrin, Bordeaux, France

REFERENCES:
- [Background] Baroud G, Nemes J, Heini P, Steffen T. Load shift of the intervertebral disc after a vertebroplasty: a finite-element study. Eur Spine J. 2003 Aug;12(4):421-6. doi: 10.1007/s00586-002-0512-9. Epub 2003 Apr 1. PMID 12687437
- [Background] Baroud G, Bohner M, Heini P, Steffen T. Injection biomechanics of bone cements used in vertebroplasty. Biomed Mater Eng. 2004;14(4):487-504. PMID 15472396
- [Background] Berlemann U, Ferguson SJ, Nolte LP, Heini PF. Adjacent vertebral failure after vertebroplasty. A biomechanical investigation. J Bone Joint Surg Br. 2002 Jul;84(5):748-52. doi: 10.1302/0301-620x.84b5.11841. PMID 12188498
- [Background] Berrington de Gonzalez A, Darby S. Risk of cancer from diagnostic X-rays: estimates for the UK and 14 other countries. Lancet. 2004 Jan 31;363(9406):345-51. doi: 10.1016/S0140-6736(04)15433-0. PMID 15070562
- [Background] Black DM, Arden NK, Palermo L, Pearson J, Cummings SR. Prevalent vertebral deformities predict hip fractures and new vertebral deformities but not wrist fractures. Study of Osteoporotic Fractures Research Group. J Bone Miner Res. 1999 May;14(5):821-8. doi: 10.1359/jbmr.1999.14.5.821. PMID 10320531
- [Background] Cooper C, Atkinson EJ, O'Fallon WM, Melton LJ 3rd. Incidence of clinically diagnosed vertebral fractures: a population-based study in Rochester, Minnesota, 1985-1989. J Bone Miner Res. 1992 Feb;7(2):221-7. doi: 10.1002/jbmr.5650070214. PMID 1570766
- [Background] Deramond H, Wright NT, Belkoff SM. Temperature elevation caused by bone cement polymerization during vertebroplasty. Bone. 1999 Aug;25(2 Suppl):17S-21S. doi: 10.1016/s8756-3282(99)00127-1. PMID 10458268
- [Background] European Prospective Osteoporosis Study (EPOS) Group; Felsenberg D, Silman AJ, Lunt M, Armbrecht G, Ismail AA, Finn JD, Cockerill WC, Banzer D, Benevolenskaya LI, Bhalla A, Bruges Armas J, Cannata JB, Cooper C, Dequeker J, Eastell R, Felsch B, Gowin W, Havelka S, Hoszowski K, Jajic I, Janott J, Johnell O, Kanis JA, Kragl G, Lopes Vaz A, Lorenc R, Lyritis G, Masaryk P, Matthis C, Miazgowski T, Parisi G, Pols HA, Poor G, Raspe HH, Reid DM, Reisinger W, Schedit-Nave C, Stepan JJ, Todd CJ, Weber K, Woolf AD, Yershova OB, Reeve J, O'Neill TW. Incidence of vertebral fracture in europe: results from the European Prospective Osteoporosis Study (EPOS). J Bone Miner Res. 2002 Apr;17(4):716-24. doi: 10.1359/jbmr.2002.17.4.716. PMID 11918229
- [Background] Evans AJ, Jensen ME, Kip KE, DeNardo AJ, Lawler GJ, Negin GA, Remley KB, Boutin SM, Dunnagan SA. Vertebral compression fractures: pain reduction and improvement in functional mobility after percutaneous polymethylmethacrylate vertebroplasty retrospective report of 245 cases. Radiology. 2003 Feb;226(2):366-72. doi: 10.1148/radiol.2262010906. PMID 12563127
- [Background] Finnern HW, Sykes DP. The hospital cost of vertebral fractures in the EU: estimates using national datasets. Osteoporos Int. 2003 Jun;14(5):429-36. doi: 10.1007/s00198-003-1395-2. Epub 2003 Apr 30. PMID 12730759
- [Background] Galibert P, Deramond H, Rosat P, Le Gars D. [Preliminary note on the treatment of vertebral angioma by percutaneous acrylic vertebroplasty]. Neurochirurgie. 1987;33(2):166-8. French. PMID 3600949
- [Background] Gauthier O, Muller R, von Stechow D, Lamy B, Weiss P, Bouler JM, Aguado E, Daculsi G. In vivo bone regeneration with injectable calcium phosphate biomaterial: a three-dimensional micro-computed tomographic, biomechanical and SEM study. Biomaterials. 2005 Sep;26(27):5444-53. doi: 10.1016/j.biomaterials.2005.01.072. PMID 15860201
- [Background] Gheduzzi S, Webb JJ, Miles AW. Mechanical characterisation of three percutaneous vertebroplasty biomaterials. J Mater Sci Mater Med. 2006 May;17(5):421-6. doi: 10.1007/s10856-006-8469-6. PMID 16688582
- [Background] Graham J, Ahn C, Hai N, Buch BD. Effect of bone density on vertebral strength and stiffness after percutaneous vertebroplasty. Spine (Phila Pa 1976). 2007 Aug 15;32(18):E505-11. doi: 10.1097/BRS.0b013e318133fc73. PMID 17700430
- [Background] Hulme PA, Krebs J, Ferguson SJ, Berlemann U. Vertebroplasty and kyphoplasty: a systematic review of 69 clinical studies. Spine (Phila Pa 1976). 2006 Aug 1;31(17):1983-2001. doi: 10.1097/01.brs.0000229254.89952.6b. PMID 16924218
- [Background] Kado DM, Duong T, Stone KL, Ensrud KE, Nevitt MC, Greendale GA, Cummings SR. Incident vertebral fractures and mortality in older women: a prospective study. Osteoporos Int. 2003 Jul;14(7):589-94. doi: 10.1007/s00198-003-1412-5. Epub 2003 Jun 24. PMID 12827222
- [Background] Kuklo TR, Polly DW, Owens BD, Zeidman SM, Chang AS, Klemme WR. Measurement of thoracic and lumbar fracture kyphosis: evaluation of intraobserver, interobserver, and technique variability. Spine (Phila Pa 1976). 2001 Jan 1;26(1):61-5; discussion 66. doi: 10.1097/00007632-200101010-00012. PMID 11148647
- [Background] Lindsay R, Silverman SL, Cooper C, Hanley DA, Barton I, Broy SB, Licata A, Benhamou L, Geusens P, Flowers K, Stracke H, Seeman E. Risk of new vertebral fracture in the year following a fracture. JAMA. 2001 Jan 17;285(3):320-3. doi: 10.1001/jama.285.3.320. PMID 11176842
- [Background] Molloy S, Riley LH 3rd, Belkoff SM. Effect of cement volume and placement on mechanical-property restoration resulting from vertebroplasty. AJNR Am J Neuroradiol. 2005 Feb;26(2):401-4. PMID 15709144
- [Background] Old JL, Calvert M. Vertebral compression fractures in the elderly. Am Fam Physician. 2004 Jan 1;69(1):111-6. PMID 14727827
- [Background] Polikeit A, Nolte LP, Ferguson SJ. The effect of cement augmentation on the load transfer in an osteoporotic functional spinal unit: finite-element analysis. Spine (Phila Pa 1976). 2003 May 15;28(10):991-6. doi: 10.1097/01.BRS.0000061987.71624.17. PMID 12768136
- [Background] Riggs BL, Melton LJ 3rd. The worldwide problem of osteoporosis: insights afforded by epidemiology. Bone. 1995 Nov;17(5 Suppl):505S-511S. doi: 10.1016/8756-3282(95)00258-4. PMID 8573428
- [Background] Ryu KS, Park CK, Kim MC, Kang JK. Dose-dependent epidural leakage of polymethylmethacrylate after percutaneous vertebroplasty in patients with osteoporotic vertebral compression fractures. J Neurosurg. 2002 Jan;96(1 Suppl):56-61. doi: 10.3171/spi.2002.96.1.0056. PMID 11795714
- [Background] Zoarski GH, Snow P, Olan WJ, Stallmeyer MJ, Dick BW, Hebel JR, De Deyne M. Percutaneous vertebroplasty for osteoporotic compression fractures: quantitative prospective evaluation of long-term outcomes. J Vasc Interv Radiol. 2002 Feb;13(2 Pt 1):139-48. doi: 10.1016/s1051-0443(07)61930-7. PMID 11830619